CLINICAL TRIAL: NCT04787211
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Human Monoclonal Antibodies, BRII-196 and BRII-198, Administered by Intravenous Infusion for the Treatment of COVID-19 Patients
Brief Title: A Study of Human Monoclonal Antibodies, BRII-196 and BRII-198
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brii Biosciences Limited (Industry)
Collaborators: TSB Therapeutics (Beijing) CO.LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRII-196-198-004
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19 phase 2; monoclonal antibody
MeSH Terms: conditions — COVID-19 | interventions — amubarvimab; romlusevimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BRII-196 and BRII-198 in adult subjects with severe COVID-19 (Experimental)
  Interventions: Drug: BRII-196 and BRII-198
- BRII-196 and BRII-198 in adult subjects with mild-moderate COVID-19 (Experimental)
  Interventions: Drug: BRII-196 and BRII-198
- Placebo in adult subjects with mild-moderate COVID-19 (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BRII-196 and BRII-198 — BRII-196 and BRII-198 given by intravenous administration
  Arms: BRII-196 and BRII-198 in adult subjects with mild-moderate COVID-19; BRII-196 and BRII-198 in adult subjects with severe COVID-19
Drug: Placebo — Placebo given by intravenous administration
  Arms: Placebo in adult subjects with mild-moderate COVID-19

SUMMARY:
The aim of this phase 2 study is to evaluate the safety and efficacy of single dose IV infusion of BRII-196 and BRII-198 given as combination therapy in patients with severe COVID-19, and mild to moderate COVID-19 and asymptomatic carrier.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 18 years, signing the informed consent.
* SARS-CoV-2 infection by PCR ≤ 7 days
* One or more of COVID-19 related symptoms or measured fever present within 48 hours prior to study entry (subjects with mild-moderate COVID-19)

Exclusion Criteria:

* Recurring COVID-19 patients
* Subjects with any unstable conditions, a history of significant hypersensitivity, or known allergy to components of the investigational agent
* Receipt of convalescent COVID-19 plasma, SARS-CoV-2 mAb treatment, SARS-CoV-2 vaccine, or other investigational treatments prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to Day 181
Incidence of serious adverse events (SAEs) | Up to Day 181
Change from pre-dose baseline in RBC count | Day 29
Change from pre-dose baseline in WBC count | Day 29
Change from pre-dose baseline in Platelets count | Day 29
Change from pre-dose baseline in Hemoglobin result | Day 29
Change from pre-dose baseline in Creatine kinase result | Day 29
Change from pre-dose baseline in Alanine aminotransferase (ALT) result | Day 29
Time-weighted average changes in SARSCoV-2 RNA levels in nasopharyngeal swabs from baseline to Day 8 | Day 8

SECONDARY OUTCOMES:
Duration of COVID-19 related symptoms through Day 29 among subjects with mild-moderate COVID-19 | up to Day 29
Proportion of subjects who have mild-moderate COVID-19 and develop severe COVID-19 after randomization | up to 26 weeks
Assessment of PK parameters (Group A and B): maximum serum concentration observed (Cmax) | up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, MD, Study Chair — Leading Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University; Fujie Zhang, MD, Principal Investigator — Co-Study Chair, Beijing Ditan Hospital Capital Medical University; Jing Yuan, MD, Principal Investigator — Site-PI, The Third People's Hospital of Shenzhen; Xilong Deng, MMS, Principal Investigator — Site-PI, Guangzhou Eighth Hospital, Guangzhou Medical University; Yao Zhang, MD, Study Director — TSB Therapeutics (Beijing) CO.LTD; Xingxiang Xu, MD, Principal Investigator — Site-PI, Subei People's Hospital of Jiangsu province; Xinping Yang, BMED, Principal Investigator — Site-PI, Yunnan Provincial Infectious Disease Hospital
Locations (6):
- China (6):
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Guangzhou Eighth Hospital, Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - Yunnan Provincial Infectious Disease Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343